CLINICAL TRIAL: NCT01955707
Title: A Multicenter, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group Study to Evaluate the Safety and Efficacy of Intravenous Natalizumab (BG00002) on Reducing Infarct Volume in Acute Ischemic Stroke
Brief Title: Effect of Natalizumab on Infarct Volume in Acute Ischemic Stroke
Acronym: ACTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101SK201; EUDRA CT NO: 2013-001514-15
Record Dates: First submitted 2013-09-30; First posted 2013-10-07 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-05

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Natalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- natalizumab (Experimental): 300 mg single intravenous (IV) injection
  Interventions: Drug: natalizumab
- Placebo (Placebo Comparator): A single IV dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: natalizumab — Administered as described in the treatment arm
  Other Names: Tysabri; BG00002
  Arms: natalizumab
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine whether one 300 mg dose of intravenous (IV) natalizumab reduces change in infarct volume from Baseline to Day 5 on magnetic resonance imaging (MRI) in participants with acute ischemic stroke when given at ≤6 hours or at >6 to ≤9 hours from when they were last known normal (LKN).

The secondary objectives of this study in this study population are as follows: to assess the efficacy of natalizumab on change in infarct volume from Baseline to Day 30; to assess efficacy of natalizumab on change in infarct volume from 24 hours to Day 5 and Day 30; to assess the efficacy of natalizumab on clinical measures of stroke outcome; to assess the safety of natalizumab in participants with acute ischemic stroke.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of acute ischemic stroke.
* Score of ≥6 points on the National Institute of Health Stroke Scale (NIHSS) at Screening.
* At least 1 acute infarct with largest diameter of more than 2 cm on Baseline brain diffusion-weighted imaging (DWI).
* Participants who have received reperfusion therapy may be eligible to participate but must meet all eligibility criteria and perform the Baseline study magnetic resonance imaging (MRI) after reperfusion therapy has been completed.
* Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for at least 3 months after their dose of study treatment.

Key Exclusion Criteria:

* Presence of any intracranial hemorrhage (ICH) on head computed tomography (CT) or non-petechial ICH on screening MRI.
* Stroke isolated to the brainstem.
* Presence of coma
* Expected to die OR unable to be evaluated within 5 days.
* Hypotension requiring the use of intravenous (IV) vasopressor support or systolic blood pressure <90 mmHg at the time of randomization.
* Known prior treatment with natalizumab.
* Immunocompromised subjects, as determined by the Investigator.
* History of progressive multifocal leukoencephalopathy (PML).
* Contraindications to MRI, e.g., implanted pacemaker or other contraindicated implanted metal devices, history of or risk for side effects from gadolinium, or claustrophobia that cannot be medically managed.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (46):
- United States (19):
  - Research Site, San Diego, California
  - Research Site, Gainesville, Florida
  - Research Site, Kansas City, Kansas
  - Research Site, Boston, Massachusetts
  - Research Site, Golden Valley, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Lake Success, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Tualatin, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Milwaukee, Wisconsin
- Germany (16):
  - Research Site, Altenburg
  - Research Site, Bad Neustadt an der Saale
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Düsseldorf
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Idar-Oberstein
  - Research Site, Leipzig
  - Research Site, Ludwigshafen
  - Research Site, Mannheim
  - Research Site, Trier
  - Research Site, Tübingen
  - Research Site, Ulm
- Spain (11):
  - Research Site, Albacete
  - Research Site, Badalona
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid

REFERENCES:
- [Derived] Elkins J, Veltkamp R, Montaner J, Johnston SC, Singhal AB, Becker K, Lansberg MG, Tang W, Chang I, Muralidharan K, Gheuens S, Mehta L, Elkind MSV. Safety and efficacy of natalizumab in patients with acute ischaemic stroke (ACTION): a randomised, placebo-controlled, double-blind phase 2 trial. Lancet Neurol. 2017 Mar;16(3):217-226. doi: 10.1016/S1474-4422(16)30357-X. Epub 2017 Feb 15. PMID 28229893

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: A single intravenous (IV) injection of placebo
- Natalizumab: 300 mg single IV injection of natalizumab
Period: Overall Study
Arm/Group | Placebo | Natalizumab
Started | 82 | 79
Withdrew Prior to Dosing | 0 | 1
Dosed | 82 | 78
Received Total Volume of Study Drug | 82 | 77
Completed | 62 | 57
Not Completed | 20 | 22
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Death | 13 | 14
Not completed — Other | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: A single IV injection of placebo
- Total: Total of all reporting groups
Arm/Group | Placebo | Natalizumab | Total
Number analyzed (Participants) | 82 | 79 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (11.83) | 70.3 (13.34) | 71.0 (12.57)
Age, Customized [Number; unit: participants]
  </= 39 years | 2 | 3 | 5
  40 to 59 years | 13 | 11 | 24
  60 to 79 years | 41 | 45 | 86
  >/= 80 years | 26 | 20 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | 72
  Male | 48 | 41 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change in Infarct Volume From Baseline (Diffusion-Weighted Imaging [DWI]) to Day 5 (Fluid-Attenuated Inversion Recovery [FLAIR])
Description: Relative growth of infarct volume from Baseline (relative growth = FLAIR at Day 5 divided by Baseline DWI). Geometric mean calculated as the exponential of the mean log relative growth.
Time Frame: Baseline, Day 5
Population: Modified intention to treat (all participants who were randomized and received the entire infusion of study treatment) with assessments at both time points.
Measure: Geometric Mean (Inter-Quartile Range); unit: mL
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 73 | 69
mL | 2.17 [1.60 to 3.17] | 2.37 [1.51 to 2.91]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab; Treatment contrasts derived from a repeated measures mixed effects model modeling log relative growth relative to baseline using an autoregressive variance-covariance matrix structure. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, and tissue plasminogen activator (tPA) use; Test type: Superiority or Other; adjusted mean difference (log-scale) = 0.08, 90% CI 2-sided [-0.09 to 0.26]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab; Test type: Superiority or Other; p = 0.779, repeated measures mixed effects model — one-sided p-value; ratio of relative growth = 1.09, 90% CI 2-sided [0.91 to 1.30] — Adjusted mean (log-scale) back-transformed to the original scale as the estimated ratio of natalizumab to placebo. 90% confidence interval (log-scale) back-transformed to the original scale and reflect the interval around the ratio

2. Secondary Outcome: Change in Infarct Volume From Baseline (DWI) to 24 Hours (FLAIR)
Description: Relative growth of infarct volume from Baseline (relative growth = FLAIR at 24 hours divided by Baseline DWI). Geometric mean calculated as the exponential of the mean log relative growth.
Time Frame: Baseline, 24 hrs
Population: as for outcome 1
Measure: Geometric Mean (Inter-Quartile Range); unit: mL
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 74 | 69
mL | 1.73 [1.33 to 2.15] | 1.95 [1.36 to 2.20]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab; Treatment contrasts derived from a repeated measures mixed effects model modeling log relative growth relative to baseline using an autoregressive variance-covariance matrix structure. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, and tPA use; Test type: Superiority or Other; adjusted mean difference (log-scale) = 0.09, 90% CI 2-sided [-0.09 to 0.27]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab; Test type: Superiority or Other; p = 0.797, repeated measures mixed effects model — one-sided p-value; ratio of relative growth = 1.09, 90% CI 2-sided [0.92 to 1.31] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Change in Infarct Volume From Baseline (DWI) to Day 30 (FLAIR)
Description: Relative growth of infarct volume from Baseline (relative growth = FLAIR at Day 30 divided by Baseline DWI). Geometric mean calculated as the exponential of the mean log relative growth.
Time Frame: Baseline, Day 30
Population: as for outcome 1
Measure: Geometric Mean (Inter-Quartile Range); unit: mL
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 66 | 55
mL | 1.27 [0.90 to 1.88] | 1.25 [0.78 to 1.93]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Adjusted mean difference (log-scale) = 0.05, 90% CI 2-sided [-0.13 to 0.24]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab; Test type: Superiority or Other; p = 0.684, repeated measures mixed effects model — one-sided p-value; ratio of relative growth = 1.05, 90% CI 2-sided [0.88 to 1.27] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Change in Infarct Volume From 24 Hours (FLAIR) to Day 5 (FLAIR)
Description: Relative growth of infarct volume from 24 hours (relative growth = FLAIR at Day 5 divided by FLAIR at 24 hours). Geometric mean calculated as the exponential of the mean log relative growth.
Time Frame: 24 hours, Day 5
Population: as for outcome 1
Measure: Geometric Mean (Inter-Quartile Range); unit: mL
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 70 | 65
mL | 1.27 [1.11 to 1.37] | 1.25 [1.11 to 1.42]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab; Treatment contrasts derived from a repeated measures mixed effects model modeling log relative growth relative to 24 hours using an autoregressive variance-covariance matrix structure. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, and tPA use; Test type: Superiority or Other; Adjusted mean difference (log-scale) = -0.00, 90% CI 2-sided [-0.12 to 0.11]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab; Test type: Superiority or Other; p = 0.487, repeated measures mixed effects model — one-sided p-value; ratio of relative growth = 1.00, 90% CI 2-sided [0.89 to 1.12] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Change in Infarct Volume From 24 Hours (FLAIR) to Day 30 (FLAIR)
Description: Relative growth in infarct volume from Baseline (relative growth = FLAIR Day 30 divided by FLAIR at 24 hours ). Geometric mean calculated as the exponential of the mean log relative growth.
Time Frame: 24 hours, Day 30
Population: as for outcome 1
Measure: Geometric Mean (Inter-Quartile Range); unit: mL
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 62 | 53
mL | 0.75 [0.62 to 1.03] | 0.72 [0.56 to 1.09]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Adjusted mean difference (log-scale) = -0.02, 90% CI 2-sided [-0.14 to 0.10]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab; Test type: Superiority or Other; p = 0.402, repeated measures mixed effects model — one-sided p-value; ratio of relative growth = 0.98, 90% CI 2-sided [0.87 to 1.11] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Change in Infarct Volume From Day 5 (FLAIR) to Day 30 (FLAIR)
Description: Relative growth of infarct volume from Day 5 (relative growth = FLAIR at Day 30 divided by FLAIR at Day 5). Geometric mean calculated as the exponential of the mean log relative growth.
Time Frame: Day 5, Day 30
Population: as for outcome 1
Measure: Geometric Mean (Inter-Quartile Range); unit: mL
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 64 | 54
mL | 0.60 [0.52 to 0.79] | 0.59 [0.42 to 0.81]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab; Treatment contrasts derived from a repeated measures mixed effects model modeling log relative growth relative to Day 5 using an autoregressive variance-covariance matrix structure. The model adjusts for for treatment, log baseline DWI volume, treatment time window, and tPA use; Test type: Superiority or Other; Adjusted mean difference (log-scale) = -0.02, 90% CI 2-sided [-0.18 to 0.13]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab; Test type: Superiority or Other; p = 0.394, repeated measures mixed effects model — one-sided p-value; ratio of relative growth = 0.98, 90% CI 2-sided [0.84 to 1.14] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Change in National Institute of Health Stroke Scale (NIHSS) Score From Baseline to 24 Hours, Day 5, Day 30, and Day 90
Description: The NIHSS is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Scores for the NIHSS range from 0 to 42, with 0 representing no symptoms and 42 representing death.
Time Frame: Baseline, 24 hours, Day 5, Day 30, Day 90
Population: Modified intention to treat (all participants who were randomized and received the entire infusion of study treatment); n=participants with assessments at Baseline and given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 82 | 77
units on a scale
  Change at 24 hours; n=82, 77 | -1.5 (3.96) | -1.5 (5.10)
  Change at Day 5; n=79, 72 | -3.3 (5.31) | -2.1 (6.24)
  Change at Day 30; n=73, 62 | -5.7 (5.22) | -4.9 (5.73)
  Change at Day 90; n=62, 56 | -7.3 (3.95) | -6.8 (5.78)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab; Analysis of NIHSS score and change from Baseline at 24 hours. The repeated measures mixed effects model is modeling absolute change in NIHSS score relative to baseline and using an autoregressive variance-covariance matrix. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, tPA use, baseline NIHSS score and location of stroke; Test type: Superiority or Other; p = 0.427, repeated measures mixed effects model — one-sided p-value; adjusted mean change from baseline = -0.25, 90% CI 2-sided [-2.48 to 1.98]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab; Analysis of NIHSS score and change from Baseline at Day 5. The repeated measures mixed effects model is modeling absolute change in NIHSS score relative to baseline and using an autoregressive variance-covariance matrix. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, tPA use, baseline NIHSS score and location of stroke; Test type: Superiority or Other; p = 0.896, repeated measures mixed effects model — one-sided p-value; adjusted mean change from baseline = 1.71, 90% CI 2-sided [-0.52 to 3.94]
Statistical Analysis 3: Comparison: Placebo vs Natalizumab; Analysis of NIHSS score and change from Baseline at Day 30. The repeated measures mixed effects model is modeling absolute change in NIHSS score relative to baseline and using an autoregressive variance-covariance matrix. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, tPA use, baseline NIHSS score and location of stroke; Test type: Superiority or Other; p = 0.989, repeated measures mixed effects model — one-sided p-value; adjusted mean change from baseline = 3.15, 90% CI 2-sided [0.89 to 5.40]
Statistical Analysis 4: Comparison: Placebo vs Natalizumab; Analysis of NIHSS score and change from Baseline at Day 90. The repeated measures mixed effects model is modeling absolute change in NIHSS score relative to baseline and using an autoregressive variance-covariance matrix. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, tPA use, baseline NIHSS score and location of stroke; Test type: Superiority or Other; p = 0.915, repeated measures mixed effects model — one-sided p-value; adjusted mean change from baseline = 1.93, 90% CI 2-sided [-0.38 to 4.25]

8. Secondary Outcome: Modified Rankin Scale (mRS) Distribution at Day 5, Day 30, and Day 90
Description: The mRS measures independence, rather than neurologic function, with specific tasks pre- and post-stroke, respectively. The scale consists of 7 grades, from 0 to 6, with 0 corresponding to no symptoms and 6 corresponding to death. The distribution of mRS scores was summarized at each timepoint. An excellent outcome on the mRS was defined as a score of 0 or 1, while a good outcome was defined as a score of 0, 1, or 2.
Time Frame: Day 5, Day 30, and Day 90
Population: Modified intention to treat (all participants who were randomized and received the entire infusion of study treatment), using imputed data; n=number of participants with an assessment at given time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 82 | 77
participants
  Day 5: Score 0; n=82, 76 | 0 | 2
  Day 5: Score 1; n=82, 76 | 3 | 2
  Day 5: Score 2; n=82, 76 | 10 | 11
  Day 5: Score 3; n=82, 76 | 13 | 11
  Day 5: Score 4; n=82, 76 | 25 | 16
  Day 5: Score 5; n=82, 76 | 29 | 31
  Day 5: Score 6; n=82, 76 | 2 | 3
  Day 30: Score 0; n=81, 72 | 0 | 5
  Day 30: Score 1; n=81, 72 | 7 | 8
  Day 30: Score 2; n=81, 72 | 14 | 8
  Day 30: Score 3; n=81, 72 | 17 | 17
  Day 30: Score 4; n=81, 72 | 22 | 14
  Day 30: Score 5; n=81, 72 | 13 | 11
  Day 30: Score 6; n=81, 72 | 8 | 9
  Day 90: Score 0; n=78, 72 | 4 | 8
  Day 90: Score 1; n=78, 72 | 12 | 10
  Day 90: Score 2; n=78, 72 | 12 | 10
  Day 90: Score 3; n=78, 72 | 15 | 13
  Day 90: Score 4; n=78, 72 | 14 | 11
  Day 90: Score 5; n=78, 72 | 8 | 6
  Day 90: Score 6; n=78, 72 | 13 | 14
Statistical Analysis 1: Comparison: Placebo vs Natalizumab; Analysis of distribution of mRS scores at Day 5. Odds ratio from a proportional-odds logistic regression model assuming a common odds ratio across all cut points of the mRS score. Covariates include baseline DWI volume (< median vs >= median), treatment time window, location of stroke abnormality (cortical/subcortical), and tPA use (yes/no); Test type: Superiority or Other; p = 0.564, Van Elteren's test — One sided p-value based on Van Elteren's test, adjusting for baseline DWI volume (< median vs >= median), treatment time window, location of stroke abnormality (cortical/subcortical), and tPA use (yes/no); Odds Ratio (OR) = 0.89, 90% CI 2-sided [0.55 to 1.45]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab; Analysis of distribution of mRS scores at Day 30. Odds ratio from a proportional-odds logistic regression model assuming a common odds ratio across all cut points of the mRS score. Covariates include baseline DWI volume (< median vs >= median), treatment time window, location of stroke abnormality (cortical/subcortical), and tPA use (yes/no); Test type: Superiority or Other; p = 0.077, Van Elteren's test — One-sided p-value based on Van Elteren's test, adjusting for baseline DWI volume (< median vs >= median), treatment time window, location of stroke abnormality (cortical/subcortical), and tPA use (yes/no); Odds Ratio (OR) = 1.30, 90% CI 2-sided [0.80 to 2.10]
Statistical Analysis 3: Comparison: Placebo vs Natalizumab; Analysis of the distribution of mRS scores at Day 90. Odds ratio from a proportional-odds logistic regression model assuming a common odds ratio across all cut points of the mRS score. Covariates include baseline DWI volume (< median vs >= median), treatment time window, location of stroke abnormality (cortical/subcortical), and tPA use (yes/no); Test type: Superiority or Other; p = 0.243, Van Elteren's test — One -sided p-value based on Van Elteren's test, adjusting for baseline DWI volume (< median vs >= median), treatment time window, location of stroke abnormality (cortical/subcortical), and tPA use (yes/no); Odds Ratio (OR) = 1.15, 90% CI 2-sided [0.71 to 1.86]

9. Secondary Outcome: Barthel Index at Day 5, Day 30, and Day 90
Description: The Barthel Index consists of 10 items that measure a person's daily functioning, specifically the activities of daily living and mobility, and can be used to determine a baseline level of functioning and to monitor change in activities of daily living over time. The scores for each of the items are summed to create a total score up to a potential of 100, with higher scores representing a greater level of independence.
Time Frame: Day 5, Day 30, and Day 90
Population: Modified intention to treat (all participants who were randomized and received the entire infusion of study treatment); n=participants with assessment at given time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 82 | 77
units on a scale
  Day 5; n=78, 73 | 35.0 [0 to 100] | 30.0 [0 to 100]
  Day 30; n=73, 60 | 70.0 [0 to 100] | 80.0 [0 to 100]
  Day 90; n=61, 55 | 80.0 [0 to 100] | 95.0 [0 to 100]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab; Analysis of Barthel Index at Day 5. The repeated measures mixed effects model is modeling Barthel Index using an autoregressive variance-covariance matrix. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, tPA use, and location of stroke; Test type: Superiority or Other; p = 0.455, repeated measures mixed effects model — one-sided p-value; Adjusted mean = 0.68, 90% CI 2-sided [-9.19 to 10.56]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab; Analysis of Barthel Index at Day 30. The repeated measures mixed effects model is modeling Barthel Index using an autoregressive variance-covariance matrix. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, tPA use, and location of stroke; Test type: Superiority or Other; p = 0.420, repeated measures mixed effects model — one-sided p-value; Adjusted mean = 1.21, 90% CI 2-sided [-8.76 to 11.19]
Statistical Analysis 3: Comparison: Placebo vs Natalizumab; Analysis of Barthel Index at Day 90/Final Visit. The repeated measures mixed effects model is modeling Barthel Index using an autoregressive variance-covariance matrix. The model adjusts for treatment, time, treatment by time, log baseline DWI volume, treatment time window, tPA use, and location of stroke; Test type: Superiority or Other; p = 0.283, repeated measures mixed effects model; Adjusted mean = 3.56, 90% CI 2-sided [-6.64 to 13.75]

10. Secondary Outcome: Number of Participants Who Experience Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence that does not necessarily have a causal relationship with this treatment. SAE: any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect; any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above. Events were categorized as severe, moderate, or mild, and related or not related to study treatment.
Time Frame: Up to Day 90 ± 5 days
Population: Safety population (all participants who were randomized and received any portion of the infusion of study treatment).
Measure: Number; unit: participants
Arm/Group | Placebo | Natalizumab
Number analyzed (Participants) | 82 | 78
participants
  Participants with an event | 81 | 77
  Participants with a moderate or severe event | 60 | 53
  Participants with a severe event | 27 | 22
  Participants with a related event | 7 | 6
  Participants with a serious event | 38 | 36
  Participants discontinuing due to an event | 0 | 0
  Participants withdrawing from study due to event | 2 | 1

ADVERSE EVENTS:
Time Frame: From informed consent (SAE) or initiation of study drug (AE) until Final Visit Day 90 ± 5 days or early termination follow-up.
Arm/Group | Placebo | Natalizumab
Serious Adverse Events (participants affected / at risk) | 38/82 | 36/78
Other Adverse Events (participants affected / at risk) | 75/82 | 68/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=82) | Natalizumab (N=78)
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Death (General disorders) | 0 | 1
Device dislocation (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Respiratory tract infection (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basilar artery thrombosis (Nervous system disorders) | 1 | 0
Brain midline shift (Nervous system disorders) | 1 | 1
Brain oedema (Nervous system disorders) | 2 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 3
Cerebral infarction (Nervous system disorders) | 2 | 4
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Convulsion (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 0 | 1
Dementia alzheimer's type (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Generalised non-convulsive epilepsy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 3 | 4
Headache (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 2 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Stroke in evolution (Nervous system disorders) | 0 | 2
Subdural hygroma (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Endarterectomy (Surgical and medical procedures) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=82) | Natalizumab (N=78)
Anaemia (Blood and lymphatic system disorders) | 4 | 8
Atrial fibrillation (Cardiac disorders) | 10 | 7
Bradycardia (Cardiac disorders) | 5 | 1
Tachycardia (Cardiac disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 23 | 24
Nausea (Gastrointestinal disorders) | 11 | 9
Vomiting (Gastrointestinal disorders) | 15 | 5
Pain (General disorders) | 6 | 9
Pyrexia (General disorders) | 26 | 32
Pneumonia (Infections and infestations) | 6 | 10
Respiratory tract infection (Infections and infestations) | 9 | 4
Urinary tract infection (Infections and infestations) | 13 | 19
Fall (Injury, poisoning and procedural complications) | 4 | 8
Alanine aminotransferase increased (Investigations) | 1 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 4
Gamma-glutamyltransferase increased (Investigations) | 5 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4
Brain oedema (Nervous system disorders) | 3 | 6
Cerebral haemorrhage (Nervous system disorders) | 0 | 4
Haemorrhagic transformation stroke (Nervous system disorders) | 21 | 18
Headache (Nervous system disorders) | 19 | 13
Neurological decompensation (Nervous system disorders) | 2 | 4
Somnolence (Nervous system disorders) | 3 | 4
Agitation (Psychiatric disorders) | 3 | 11
Anxiety (Psychiatric disorders) | 1 | 6
Depression (Psychiatric disorders) | 13 | 5
Insomnia (Psychiatric disorders) | 13 | 7
Post stroke depression (Psychiatric disorders) | 2 | 4
Sleep disorder (Psychiatric disorders) | 7 | 8
Urinary retention (Renal and urinary disorders) | 6 | 5
Hypertension (Vascular disorders) | 10 | 15
Hypotension (Vascular disorders) | 12 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.